CLINICAL TRIAL: NCT01159223
Title: A Multicenter Randomized Study to Compare the Efficacy and Safety of Lower Dose Atazanavir /Ritonavir (ATV/r 200/100 OD) Versus Standard Dose (ATV/r 300/100 mg OD) in Combination With 2NRTIs in Well Virology Suppressed HIV-infected Adults
Brief Title: Low Dose Atazanavir/r Versus Standard Dose Atazanavir/r (LASA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Kirby Institute (Other Government); National Health Security Office, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIV - NAT 110
Record Dates: First submitted 2010-06-04; First posted 2010-07-09 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: HIV Infections
Keywords: atazanavir / ritonavir; low dose; noninferiority; safety and efficacy; efficacy and safety of lower dose atazanavir/ritonavir in suppressed HIV-infected adults
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ATV/r 200 mg/100 mg OD
  Interventions: Drug: ATV/r
- 2 (Experimental): ATV/r 300 mg/100 mg OD
  Interventions: Drug: ATV/r

INTERVENTIONS:
Drug: ATV/r — All participants will be randomized to take ATV/r 200 mg/100 mg OD or ATV/r 300/100 mg OD. NRTIs background regimens will remain unchanged if possible. NRTIs background may include zidovudine/lamivudine, zidovudine plus ddI, ddI plus lamivudine, tenofovir plus lamivudine, tenofovir/emtricitabine, zidovudine plus tenofovir. NRTI backbone could be switched or modified due to toxicity or intolerance

SUMMARY:
This study will compare the efficacy and safety of ATV/r at either 200/100 mg or 300/100mg given daily in Thai patients in combination with 2NRTIs.

DETAILED DESCRIPTION:
To demonstrate non-inferiority of treatment with atazanavir/ritonavir (ATV/r) 200/100 mg once daily (OD) compared to the control group (ATV/r 300/100 mg OD) in regards to the proportion of virologic responders (plasma HIV RNA < 200 copies/mL) at 48 weeks in ARV-experienced HIV-1 infected subjects.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infected adults aged more than or equal to 18 years
2. Received ritonavir boosted PI-based HAART for >3 months prior screening visit
3. History of HIV RNA < 50 copies/ml within 12 months prior to screening visit
4. HIV-RNA < 50 copies/ml at screening visit
5. Signed written informed consent

Exclusion Criteria:

1. Active AIDS-defining disease or active opportunistic infection
2. History of virological failure (plasma HIV-RNA ≥1,000 copies/ml) while using any ritonavir boosted PI-based HAART
3. Pregnancy or lactation at screening visit
4. Relevant history or current conditions or illnesses that might interfere with drug absorption, distribution, metabolism or excretion e.g. chronic diarrhea, malabsorption
5. Use of concomitant medication that may interfere with the pharmacokinetics of the study drugs e.g. rifampicin, proton pump inhibitor
6. History of sensitivity/idiosyncrasy to the drug or chemically related compounds which may be employed in the study
7. ALT ≥200 IU/L at screening visit
8. Creatinine clearance < 60 c.c. per min by Cockroft-Gault formula at screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
noninferiority | Dec. 2013
  ATV/r 200/100 mg will be judged to be non-inferior to ATV 300/100mg if the lower limit of the 95% confidence interval for the difference in proportion of patients with virological response between the two groups does not exceed -10%

SECONDARY OUTCOMES:
viral load | DEc. 2013
  A secondary efficacy analysis will explore the impact of changing the lower limit of detection of viral load to <50 copies/mL
serious adverse events | Dec. 2013
  Changes in HDL, LDL, cholesterol, triglycerides and bilirubin, or having grade 3 and 4 laboratory adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — HIV-NAT, The Thai Red Cross AIDS Research Centre (TRCARC), and Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand
Locations (10):
- Thailand (10):
  - Chiang Rai Regional Hospital, Chiang Rai, Changwat Chiang Rai
  - ChonBuri Hospital, Chon Buri, Changwat Chon Buri
  - Khon Kaen University, Khon Kaen, Changwat Khon Kaen
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi, Changwat Nonthaburi
  - Sanpathong Hospital, Sanpathong, Chiang Mai
  - HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok
  - BMA Medical College and Vajira Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Taksin hospital, Bangkok
  - Khon Kaen Hospital, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
study protocol available at www.hivnat.org

REFERENCES:
- [Result] Bunupuradah T, Kiertiburanakul S, Avihingsanon A, Chetchotisakd P, Techapornroong M, Leerattanapetch N, Kantipong P, Bowonwatanuwong C, Banchongkit S, Klinbuayaem V, Mekviwattanawong S, Nimitvilai S, Jirajariyavej S, Prasithsirikul W, Munsakul W, Bhakeecheep S, Chaivooth S, Phanuphak P, Cooper DA, Apornpong T, Kerr SJ, Emery S, Ruxrungtham K; LASA Study Group. Low-dose versus standard-dose ritonavir-boosted atazanavir in virologically suppressed Thai adults with HIV (LASA): a randomised, open-label, non-inferiority trial. Lancet HIV. 2016 Aug;3(8):e343-e350. doi: 10.1016/S2352-3018(16)30010-8. Epub 2016 May 24. PMID 27470026
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org